CLINICAL TRIAL: NCT02056639
Title: Prevention of Preterm Birth With a Pessary in Twin Gestations
Acronym: PoPPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 819122
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Premature Birth; Short Cervix
Keywords: Premature birth; Premature delivery; Short cervix; Pessary
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pessary (Experimental): Use of the Bioteque cup pessary. Pessary will be placed between 18 and 27 6/7 weeks gestation, and will be removed during the 36th week of pregnancy (or earlier if indicated)
  Interventions: Device: Bioteque cup pessary
- No pessary (No Intervention): No pessary will be used. Subjects will receive standard obstetrical management

INTERVENTIONS:
Device: Bioteque cup pessary
  Arms: Pessary

SUMMARY:
Preterm birth (PTB) is a major health problem and contributes to more than 50% of the overall perinatal mortality. Twins are at increased risk for PTB. The number of twins births has risen substantially due to the increased use of assisted reproductive technology. The rate of twin births in the United States rose from 18.9 to 32.2 per 100 live births between 1980 and 2004. The increased rate of PTB in twins is associated with increased morbidity and mortality rates. Almost one in four very low birth-weight infants (below 1500 g) born in the United States are twins, as are one in six infants who die in the first month of life. Cervical shortening is a risk factor for PTB. Transvaginal ultrasound measurement of cervical length is a reliable screening test for prediction of PTB. There is currently no effective treatment to decrease the incidence of PTB in women with twin gestations, but there is some evidence that the use of a cervical pessary in women with a short cervix has promise. If effective this approach would be particularly appealing because of the wide availability of pessaries, ease of use, and low cost. Unfortunately, existing studies are inadequate to confirm effectiveness; a well designed, properly powered, prospective randomized trial is warranted prior to widespread implementation in clinical practice. We propose such a trial to study the effectiveness of the pessary in decreasing the incidence of PTB in an inner city Philadelphia population.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Twin pregnancy (limits the participants to female gender)
* Short cervical length (less than or equal to 30 mm) on second trimester ultrasound at 18-27 6/7 weeks gestation

Exclusion Criteria:

* Singleton or higher order than twins multiple gestation
* Monoamniotic twins
* Twin twin transfusion syndrome
* Ruptured membranes
* Lethal fetal structural anomaly
* Fetal chromosomal abnormality
* Cerclage in place (or planned placement)
* Vaginal bleeding
* Suspicion of chorioamnionitis
* Ballooning of membranes outside the cervix into the vagina
* Painful regular uterine contractions
* Labor
* Placenta previa

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Dugoff, MD, Principal Investigator — University of Pennsylvania; Vincenzo Berghella, Principal Investigator — Thomas Jefferson University; Jack Ludmir, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Pessary: Use of the Bioteque cup pessary. Pessary will be placed between 18 and 27 6/7 weeks gestation, and will be removed during the 36th week of pregnancy (or earlier if indicated)
  Bioteque cup pessary
Period: Overall Study
Arm/Group | Pessary | No Pessary
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pessary | No Pessary | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Preterm Delivery
Time Frame: Less than 34 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 23 | 23
Participants | 9 | 8

2. Secondary Outcome: Average Birth Weight of Babies in Each Group
Description: The birth weight of babies is the pessary group and no pessary group were recorded and analyzed for comparison.
Time Frame: Time of delivery
Measure: Mean (Full Range); unit: grams
Groups:
- Pessary: A biotec. pessary will be placed in subjects.
- No Pessary: No pressary will be inserted and subjects will follow standard of care.
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 23 | 23
grams | 2190 [1115 to 2540] | 2220 [1864 to 2583]

3. Secondary Outcome: Spontaneous Preterm Birth Rates
Time Frame: Less than 37 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 23 | 23
Participants | 12 | 12

4. Secondary Outcome: Number of Participants That Experienced Neonatal Death
Description: Number of participants that experienced neonatal deaths that occurred in each group following birth was recorded and analyzed.
Time Frame: Between birth and 28 days of age
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 23 | 23
Participants | 4 | 3

5. Secondary Outcome: Number of Subjects Experiencing Chorioamnionitis
Description: Chorioamnionitis was recorded and analyzed for participants in each group.
Time Frame: Time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Pessary | No Pessary
Number analyzed (Participants) | 23 | 23
Participants | 3 | 0

ADVERSE EVENTS:
Arm/Group | Pessary | No Pessary
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 3/23 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pessary (N=23) | No Pessary (N=23)
UTI (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitation of our study was the fact that it was stopped before planned enrollment was complete, which resulted in a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No